CLINICAL TRIAL: NCT04484467
Title: Efficacy and Safety of a Food Supplement With Standardized Menthol, Limonene, and Gingerol Content in Patients With Irritable Bowel Syndrome: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Efficacy and Safety of a Food Supplement With Standardized Menthol, Limonene, and Gingerol Content in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Stare Budgetary Scientific Institution, Mental Health Research Center (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other); RML INVEST, Torkhovsky passage 10, Tula, Russian Federation (Unknown)
Responsible Party: Principal Investigator, Allan G. Beniashvilia, Senior research fellow, PHD, Federal Stare Budgetary Scientific Institution, Mental Health Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 418 dated 01/31/2018
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome With Constipation; Irritable Bowel Syndrome Mixed
Keywords: Functional dyspepsia
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Dietary Supplements; Limonene; ginger extract

STUDY DESIGN:
Intervention Model Description: At Visit 1, all patients were randomly assigned into two groups. In the intervention group (Group 1), the supplement "Standart Zdorovya GASTRO" (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days. In the control group (Group 2), placebo (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days (Table 1). During the 30 days of the study, three outpatient visits were conducted (Visit 1 - Day 1, Visit 2 - Day 15 + 2 days, and Visit 3 - Day 30 + 2 days).
Who Masked: Participant, Investigator
Masking Description: Using a random number generator, 56 patients with IBS or IBS/FD were randomly assigned to either the intervention group (28 individuals) or control group (28 individuals).
  Researchers and patients were not informed who received a supplement or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement Standart Zdorovya GASTRO (Experimental): In the intervention group (Group 1), the supplement "Standart Zdorovya GASTRO" (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days.
  Interventions: Dietary Supplement: Food Supplement With Standardized Menthol, Limonene, and Ginger
- Placebo (Placebo Comparator): In the control group (Group 2), placebo (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement With Standardized Menthol, Limonene, and Ginger — Components of Standart Zdorovya GASTRO: Peppermint oil (40% menthol, 1.5% limonene) - 240 mg, Ginger oil (14% gingerol) - 50 mg, olive oil - 440 mg, 1 capsule, 730 mg, once a day for 30 days
  Other Names: Standart Zdorovya GASTRO
  Arms: Food supplement Standart Zdorovya GASTRO
Other: Placebo — Components of placebo Olive oil - 730 mg, 1 capsule, 730 mg, once a day for 30 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of a food supplement with standardized menthol, limonene, and gingerol content in patients with irritable bowel syndrome (IBS) or IBS/functional dyspepsia (FD).

DETAILED DESCRIPTION:
Using a random number generator, 56 patients meeting inclusion criteria with IBS or IBS/FD were randomly assigned to either the intervention group (28 individuals) or the control group (28 individuals) (Table 2). Non-functional causes for the symptoms were excluded by a detailed evaluation of the medical history, physical examination, extensive panel of blood tests, stool analysis, and colonoscopy with biopsies.

Diarrhoea-predominant IBS patients (IBS-D) and mixed bowel habits IBS patients (IBS-M) were treated with smooth muscle antispasmodics. The constipation-predominant IBS patients (IBS-C) were treated with smooth muscle antispasmodics and laxatives. IBS/FD patients were treated with smooth muscle antispasmodics and proton pump inhibitors.

At Visit 1, all patients were randomly assigned into two groups. In the intervention group (Group 1), the supplement "Standart Zdorovya GASTRO" (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days. In the control group (Group 2), placebo (1 capsule, 730 mg, once a day) was added to the standard treatment regimen for 30 days (Table 1). Researchers and patients were not informed who received a supplement or placebo. During the 30 days of the study, three outpatient visits were conducted (Visit 1 - Day 1, Visit 2 - Day 15 + 2 days, and Visit 3 - Day 30 + 2 days).

Symptom severity was assessed on each visit using "7x7" questionnaire [Ivashkin, V., Sheptulin, A., Shifrin, O., Poluektova, E., Pavlov, C., Ivashkin, K., Drozdova, A., Lyashenko, O., Korolev, A., 2019. Clinical validation of the "7 × 7" questionnaire for patients with functional gastrointestinal disorders. J. Gastroenterol. Hepatol. 34, 1042-1048. https://doi.org/10.1111/jgh.14546], on 1 and 3 visits stool samples were collected for the qualitative and quantitative composition of the intestinal microbiota based on 16S rRNA gene sequencing.

The study protocol was approved by the Ethics Committee of the Mental Health Research Center, Moscow, Russian Federation (No. 418 dated 01/31/2018) and written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* irritable bowel syndrome (IBS)
* diarrhea-predominant IBS
* constipation-predominant IBS
* mixed-type IBS
* IBS/functional dyspepsia symptoms
* Must be able to swallow tablets

Exclusion Criteria:

* organic bowel disease
* renal disease
* hepatic insufficiency,
* schizophrenia
* bipolar disorder
* epilepsy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Change in the severity of symptoms of irritable bowel syndrome (IBS) and functional dyspepsia (FD) (constipation-predominant, diarrhea-predominant, mixed-type IBS and IBS/FD) | Visit 1 - Day 1, Visit 2 - Day 15 +- 2 days, and Visit 3 - Day 30 +- 2 days
  Symptom severity was tested with a "7x7" questionnaire at each visit.

SECONDARY OUTCOMES:
Change in the number of SCFA producing bacteria | Visit 1 - Day 1, Visit 3 - Day 30 + 2 days
  The qualitative and quantitative composition of the intestinal microbiota was assessed at Visits 1 and 3 based on 16S rRNA gene sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivashkin VT, Kudryavtseva AV, Krasnov GS, Poluektov YM, Morozova MA, Shifrin OS, Beniashvili AG, Mamieva ZA, Kovaleva AL, Ulyanin AI, Trush EA, Erlykin AG, Poluektova EA. Efficacy and safety of a food supplement with standardized menthol, limonene, and gingerol content in patients with irritable bowel syndrome: A double-blind, randomized, placebo-controlled trial. PLoS One. 2022 Jun 15;17(6):e0263880. doi: 10.1371/journal.pone.0263880. eCollection 2022. PMID 35704960